CLINICAL TRIAL: NCT05448742
Title: Novel, Biplanar, Medial Opening Wedge, Posterior Tibial Slope-reducing High Tibial Osteotomy Aided by Patient-specific Instruments, With Tibial Tuberosity Serving as Hinge Axis: Cadaveric Study Assessing Accuracy of Biplanar Correction With Various Coronal and Sagittal Amounts of Correction
Brief Title: Biplanar PSI Slope-reducing MOWHTO With Tibial Tuberosity Serving as Hinge Axis: Cadaveric Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Konrad Malinowski MD, Director of Artromedical Konrad Malinowski Clinic and Principal Investigator, Artromedical Konrad Malinowski Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1-pro-ar-2022
Record Dates: First submitted 2022-05-18; First posted 2022-07-07 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Knee Disease; Knee Osteoarthritis; Knee Injuries and Disorders
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Six cadaveric lower limbs will have biplanar PSI slope-reducing MOWHTO performed on and accuracy of biplanar correction will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm of the study (Experimental): Six cadaveric lower limbs will have biplanar PSI slope-reducing MOWHTO performed on and accuracy of biplanar correction will be assessed.
  Interventions: Device: Biplanar PSI slope-reducing MOWHTO.

INTERVENTIONS:
Device: Biplanar PSI slope-reducing MOWHTO. — High tibial osteotomy (HTO) is a widely performed procedure in case of varus knee with medial compartment osteoarthritis (OA), with medial-opening wedge version performed more often than lateral-closing wedge one. While in most cases the goal of medial-opening wedge HTO (MOWHTO) is isolated correction of coronal limb alignment, intentional or unintentional increase of posterior tibial slope (PTS) after MOWHTO can occur, however its extent is usually limited and depends on accurate hinge axis placement. One of the ideas developed to improve accuracy of hinge axis placement and accuracy of biplanar correction are Patient-Specific Instruments (PSI). Our intervention is novel, biplanar, medial-opening wedge, posterior tibial slope-reducing high tibial osteotomy aided by PSI, with tibial tuberosity serving as hinge axis.

SUMMARY:
Six cadaveric lower limbs will have PSI slope-reducing MOWHTO performed on and accuraccy of biplanar correction will be assessed.

DETAILED DESCRIPTION:
Introduction:

High tibial osteotomy (HTO) is a widely performed procedure in case of varus knee with medial compartment osteoarthritis (OA), with medial-opening wedge version performed more often than lateral-closing wedge one. While in most cases the goal of medial-opening wedge HTO (MOWHTO) is isolated correction of coronal limb alignment, unintentional increase of posterior tibial slope (PTS) after MOWHTO can occur, however its extent is usually limited. Meta-analysis by Nha et al. published in 2016 and summarizing 27 studies including 1260 MOWHTO procedures, reported mean increase of PTS by 2.02° (95% CI, 2.66° to 1.38°; P = .005). One of factors limiting the extent of PTS change both in above described unintentional circumstances and in desired biplanar corrections, can be the fact that in most cases lateral cortex of the tibia is not transected. Therefore, increase of PTS after MOWHTO was proposed to be caused by the unique anatomical characteristics of the proximal tibia such as non-perpendicular angle between anteromedial and lateral cortex. However, this phenomenon has its limitations and in cases when greater correction of PTS is required, transection of lateral tibial cortex may be necessary, as is routinely performed in osteotomies targeted at isolated PTS correction. In such cases, posterior cortex is remained intact to serve as hinge axis.

On the other hand, in some cases significant biplanar correction of both coronal and sagittal knee alignment is desired. However, transecting all three tibial cortexes increases technical difficulty of the procedure and may increase time to union and the risk of non-union. Therefore, optimal placement of hinge axis to achieve higher accuracy of desired biplanar correction is intensively studied and discussed. In general, anterolateral placement of hinge axis is established to be necessary in order to achieve both valgus correction and PTS decrease. Such biplanar correction may be desired i.e. in anterior cruciate ligament (ACL) revision cases with varus alignment, especially in cases with associated posterolateral corner (PLC) injury, as varus alignment was shown to increase stress both in ACL and PLC grafts. What is more, Won et al. have shown that as much as 19% of ACL revision cases presented with radiographic OA of Kellgren-Lawrence 2 or higher at the medial tibiofemoral joint, highlighting the potential indication for biplanar MOWHTO. Another issue faced during MOWHTO is its influence on patellar height. Multiple studies suggested the possibility of iatrogenic lowering of the patella or the patella baja after MOWHTO. However, as early as in 1979 Goutallier et al. reported that more anterior placement of hinge axis may diminish the impact of HTO on patellar height, which remains in agreement with the proposed anterolateral placement of hinge axis. Up to date, most of the studies assessing impact of hinge axis localization on biplanar correction are based on 3D models and simulations instead of cadavers of real-life procedures, with inherent limitations of that. What is more, accurate and reproducible placement of hinge axis remains technically challenging. One of the ideas developed to improve accuracy of hinge axis placement and accuracy of biplanar correction are Patient-Specific Instruments (PSI), with good results reported by multiple authors.

Therefore, the aim of this cadaveric study was to assess accuracy of biplanar correction with precisely planned increasing various coronal and sagittal amounts of correction utilizing novel, biplanar, medial-opening wedge, posterior tibial slope-reducing high tibial osteotomy aided by PSI, with tibial tuberosity serving as hinge axis. The primary hypothesis of this study was that: 1) There will be no significant differences between planned and achieved biplanar corrections neither in coronal nor sagittal planes. Secondary hypotheses were as follows: 2) Arhtrex PEEKPower HTO plates a) provide good intraoperative stabilization, b) regardless of the change of plate location there will be enough space to preserve soft tissues and no need for new plate design. c) Material used for plates construction will allow for precise evaluation in Computed tomography (CT); 3) No intraoperative fractures will occur; 4) No significant change of patellar height will occur.

Material and Methods:

Preoperative measurements:

Six fresh-frozen cadaveric lower limbs with 2/3 distal of femoral shaft and full-length leg with ankle and feet will be included in the study. CT scans encompassing full cadaveric specimen will be performed in full extension of the knee, or in maximal extension possible in given limb. Both coronal and sagittal anatomical axis will be assessed on CT scan. Femoral anatomical axis will be defined as a line connecting center of the marrow cavity at the most proximal level of femoral shaft available and the center of the knee at the level of the line tangent to the distal ends of femoral condyles. Tibial anatomical axis will be defined as a line connecting the center of the tibial articular surface in the knee and the center of the talus, similarly to the methodology of Wu Chi-Chuan. Medial proximal tibia angle (MPTA) will be defined as the angle between tibial anatomical axis and the medial tibial plateau joint line. Anatomical femorotibial angle (aFTA) will be defined as the angle between tibial anatomical axis and femoral anatomical axis. PTS will be assessed on CT scans using the methodology provided by Meier et al. and Calek et al. Due to the fact that mean intraindividual difference between PTS measured on medial tibial condyle (medial tibial posterior slope, MTPS) and lateral tibial condyle (lateral tibial posterior slope, LTPS) was reported to differ as much as 2.9 ° (range 0.0°-10.8°) or 2.6° (range 0.0°-9.5°), MTPS and LTPS will be measured separately. They will be defined as an angles between the plane perpendicular to the mechanical axis of the tibia (established using the ankle center and tibial spine) and the line tangent to the most prominent aspects of the anterior and posterior cortices of the medial and lateral compartments, respectively.

Patellar height will be assessed utilizing Insall-Salvati Index (ISI), Blackburne-Peel Index (BPI) and Caton-Deschamps Index (CDI). Two independent observers will perform the measurements separately, each of them will perform the measurements two times. Intra- and inter-reliabilities will be calculated.

CT scans will be performed on Siemens Somatom Go Top tomograph with 140kV voltage, slice thickness 0,6mm, increment 0,4mm. Two scans will be performed during each time, with tin filter and without it. Images of better quality will be chosen for measurements Surgical procedure: All specimens will undergo novel, biplanar, medial-opening wedge, posterior tibial slope-reducing high tibial osteotomy aided by PSI, with tibial tuberosity serving as hinge axis. The following corrections will be performed: group A, 3 specimens, in all cases PTS decrease by 6° and valgus correction of anatomical axis by 6°, 9° and 12°; and group B, 3 specimens, in all cases PTS decrease by 10° and valgus correction of anatomical axis by 6°, 9° and 12°. Randomization of specimens will be performed, irrespective of their native alignment, as the primary aim of this study is to assess the accuracy of planned biplanar correction. PSI will be created for every specimen by the engineer with years of practice in designing orthopaedic PSI (author J.P.). The following computer programs will be used: for creating 3D models out of DICOM files - 3D Slicer 4.11.20210226 (Brigham and Women's Hospital (BWH) & 3D Slicer contributors, 2021); for designing 3D PSI surgical guides -SolidWorks 2016 (Dassault Systèmes SolidWorks Corporation, 2016). After completion of the design, PSI surgical guides will be 3D printed in two versions: trial, not destined for medical usage - with the 3D printer Stratasys Dimension 1200es (Stratasys Ltd), from material ABS (HMF Chemical); final, destined for medical usage - with the 3D printer EOS Formiga P110 (EOS GmbH), from material PA2200 Balance 1.0 (EOS GmbH). Obtained 3D PSI surgical guides are compliant with the requirements set out in Directive 93/42/EEC concerning medical devices as well as PN-EN ISO 15223-1, EN 1041 +A1:2013, EN ISO 14971, PN-EN ISO 17664:2005 (EN ISO 17664:2004) and PN-EN ISO 10993-1:2010 (EN ISO 10993-1:2009+AC:2010).

Postoperative measurements: MPTS, LPTS, coronal alignment and patellar height will be measured postoperatively utilizing the same methodology as described preoperatively. CT scans will be performed in the same angle of knee extension as preoperatively. Postoperative CT scans will be also assessed for the presence of fractures, in accordance with higher detection rate than when utilizing plain X-ray, as reported by Sang-June Lee. Once again, two observers will perform the measurements/ assessments separately, each of them will perform the measurements two times and they will be blinded as to desired amount of correction in the given extremity. Intra- and inter-reliabilities will be calculated. Statistical analysis will be performed in Statistica 13.3 software (StatSoft/ TIBCO Software Inc, 2017).

ELIGIBILITY:
Inclusion Criteria:

Six fresh-frozen cadaveric lower limbs with 2/3 distal of femoral shaft and full-length leg with ankle and feet will be included in the study

Exclusion Criteria:

There will be no exclusion criteria for cadaveric lower limbs.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the 3D PSI device to achieve desired Medial Proximal Tibial Angle | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to achieve desired Medial Proximal Tibial Angle - measurement of preop, postop and amount of desired and performed correction on cadavers (not clinical data, measurement on cadavers)
Feasibility of the 3D PSI device to achieve desired Medial Proximal Tibial Slope | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to achieve desired Medial Proximal Tibial Slope - measurement of preop, postop and amount of desired and performed correction on cadavers (not clinical data, measurement on cadavers)
Feasibility of the 3D PSI device to achieve desired Lateral Proximal Tibial Slope | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to achieve desired Lateral Proximal Tibial Slope - measurement of preop, postop and amount of desired and performed correction on cadavers (not clinical data, measurement on cadavers)
Feasibility of the 3D PSI device to achieve desired anatomical FemoroTibial Angle | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to achieve desired anatomical FemoroTibial Angle - measurement of preop, postop and amount of desired and performed correction on cadavers (not clinical data, measurement on cadavers)

SECONDARY OUTCOMES:
Feasibility of the 3D PSI device to avoid change of anatomical Insall-Salvati Index | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to avoid change of anatomical Insall-Salvati Index - measurement of preop and postop on cadavers (not clinical data, measurement on cadavers).
  This is a scale describing patellar height with no minimal and maximal values; higher values mean higher height of patella and lower values mean lower height of patella, however it can not be simply associated with better or worse outcome.
Feasibility of the 3D PSI device to avoid change of anatomical Blackburn-Peel Index | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to avoid change of anatomical Blackburn-Peel Index - measurement of preop and postop on cadavers (not clinical data, measurement on cadavers)
  This is a scale describing patellar height with no minimal and maximal values; higher values mean higher height of patella and lower values mean lower height of patella, however it can not be simply associated with better or worse outcome.
Feasibility of the 3D PSI device to avoid change of anatomical Caton-Deschamps Index | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to avoid change of anatomical Caton-Deschamps Index - measurement of preop and postop on cadavers (not clinical data, measurement on cadavers).
  This is a scale describing patellar height with no minimal and maximal values; higher values mean higher height of patella and lower values mean lower height of patella, however it can not be simply associated with better or worse outcome.
Feasibility of the 3D PSI device to avoid intraoperative fractures | Procedures will be perfomred on cadaveric limbs on 22th June 2022 and analyzed within 6 weeks
  Feasibility of the 3D PSI device to avoid intraoperative fractures - presence of intraoperative fractures will be assessed on CT scans (not clinical data, assessment on cadavers)

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Malinowski, MD PhD, Principal Investigator — Artromedical Orthopaedic Clinic, Bełchatów, Poland
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bin SI, Kim HJ, Ahn HS, Rim DS, Lee DH. Changes in Patellar Height After Opening Wedge and Closing Wedge High Tibial Osteotomy: A Meta-analysis. Arthroscopy. 2016 Nov;32(11):2393-2400. doi: 10.1016/j.arthro.2016.06.012. Epub 2016 Aug 25. PMID 27570171
- [Background] Calek AK, Hochreiter B, Hess S, Amsler F, Leclerq V, Hirschmann MT, Behrend H. High inter- and intraindividual differences in medial and lateral posterior tibial slope are not reproduced accurately by conventional TKA alignment techniques. Knee Surg Sports Traumatol Arthrosc. 2022 Mar;30(3):882-889. doi: 10.1007/s00167-021-06477-z. Epub 2021 Feb 6. PMID 33547913
- [Background] Dejour D, Saffarini M, Demey G, Baverel L. Tibial slope correction combined with second revision ACL produces good knee stability and prevents graft rupture. Knee Surg Sports Traumatol Arthrosc. 2015 Oct;23(10):2846-52. doi: 10.1007/s00167-015-3758-6. Epub 2015 Aug 23. PMID 26298711
- [Background] Dexel J, Fritzsche H, Beyer F, Harman MK, Lutzner J. Open-wedge high tibial osteotomy: incidence of lateral cortex fractures and influence of fixation device on osteotomy healing. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):832-837. doi: 10.1007/s00167-015-3730-5. Epub 2015 Aug 8. PMID 26254088
- [Background] Donnez M, Ollivier M, Munier M, Berton P, Podgorski JP, Chabrand P, Parratte S. Are three-dimensional patient-specific cutting guides for open wedge high tibial osteotomy accurate? An in vitro study. J Orthop Surg Res. 2018 Jul 9;13(1):171. doi: 10.1186/s13018-018-0872-4. PMID 29986731
- [Background] Eliasberg CD, Hancock KJ, Swartwout E, Robichaud H, Ranawat AS. The Ideal Hinge Axis Position to Reduce Tibial Slope in Opening-Wedge High Tibial Osteotomy Includes Proximalization-Extension and Internal Rotation. Arthroscopy. 2021 May;37(5):1577-1584. doi: 10.1016/j.arthro.2020.12.203. Epub 2020 Dec 24. PMID 33359158
- [Background] Gooi SG, Chan CXY, Tan MKL, Lim AKS, Satkunanantham K, Hui JHP. Patella Height Changes Post High Tibial Osteotomy. Indian J Orthop. 2017 Sep-Oct;51(5):545-551. doi: 10.4103/ortho.IJOrtho_214_17. PMID 28966378
- [Background] Goutallier D, Delepine G, Debeyre J. [The patello-femoral joint in osteoarthritis of the knee with genu varum (author's transl)]. Rev Chir Orthop Reparatrice Appar Mot. 1979 Jan-Feb;65(1):25-31. French. PMID 156384
- [Background] Hankemeier S, Hufner T, Wang G, Kendoff D, Zeichen J, Zheng G, Krettek C. Navigated open-wedge high tibial osteotomy: advantages and disadvantages compared to the conventional technique in a cadaver study. Knee Surg Sports Traumatol Arthrosc. 2006 Oct;14(10):917-21. doi: 10.1007/s00167-006-0035-8. Epub 2006 Feb 24. PMID 16501952
- [Background] Kesmezacar H, Erginer R, Ogut T, Seyahi A, Babacan M, Tenekecioglu Y. Evaluation of patellar height and measurement methods after valgus high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2005 Oct;13(7):539-44. doi: 10.1007/s00167-004-0572-y. Epub 2005 Jan 8. PMID 15645214
- [Background] Kim HJ, Park J, Park KH, Park IH, Jang JA, Shin JY, Kyung HS. Evaluation of Accuracy of a Three-Dimensional Printed Model in Open-Wedge High Tibial Osteotomy. J Knee Surg. 2019 Sep;32(9):841-846. doi: 10.1055/s-0038-1669901. Epub 2018 Sep 6. PMID 30189435
- [Background] Klek M, Dhawan A. The Role of High Tibial Osteotomy in ACL Reconstruction in Knees with Coronal and Sagittal Plane Deformity. Curr Rev Musculoskelet Med. 2019 Dec;12(4):466-471. doi: 10.1007/s12178-019-09589-9. PMID 31760623
- [Background] Kwun JD, Kim HJ, Park J, Park IH, Kyung HS. Open wedge high tibial osteotomy using three-dimensional printed models: Experimental analysis using porcine bone. Knee. 2017 Jan;24(1):16-22. doi: 10.1016/j.knee.2016.09.026. Epub 2016 Nov 19. PMID 27876267
- [Background] Lee BH, Ha CW, Moon SW, Chang M, Kim HY, Park SH, Wang JH. Three-dimensional relationships between secondary changes and selective osteotomy parameters for biplane medial open-wedge high tibial osteotomy. Knee. 2017 Mar;24(2):362-371. doi: 10.1016/j.knee.2016.11.010. Epub 2017 Feb 4. PMID 28169100
- [Background] Lee SJ, Kim JH, Baek E, Ryu HS, Han D, Choi W. Incidence and Factors Affecting the Occurrence of Lateral Hinge Fracture After Medial Opening-Wedge High Tibial Osteotomy. Orthop J Sports Med. 2021 Oct 8;9(10):23259671211035372. doi: 10.1177/23259671211035372. eCollection 2021 Oct. PMID 34646897
- [Background] Meier M, Janssen D, Koeck FX, Thienpont E, Beckmann J, Best R. Variations in medial and lateral slope and medial proximal tibial angle. Knee Surg Sports Traumatol Arthrosc. 2021 Mar;29(3):939-946. doi: 10.1007/s00167-020-06052-y. Epub 2020 May 10. PMID 32390118
- [Background] Miao Z, Li S, Luo D, Lu Q, Liu P. The validity and accuracy of 3D-printed patient-specific instruments for high tibial osteotomy: a cadaveric study. J Orthop Surg Res. 2022 Jan 29;17(1):62. doi: 10.1186/s13018-022-02956-2. PMID 35093132
- [Background] Moon SW, Park SH, Lee BH, Oh M, Chang M, Ahn JH, Wang JH. The Effect of Hinge Position on Posterior Tibial Slope in Medial Open-Wedge High Tibial Osteotomy. Arthroscopy. 2015 Jun;31(6):1128-33. doi: 10.1016/j.arthro.2015.01.009. Epub 2015 Mar 3. PMID 25744929
- [Background] Neyret P, Zuppi G, Selmi TA (2000) Tibial deflexion osteotomy. Oper Tech Sports Med 8:61-66
- [Background] Nha KW, Kim HJ, Ahn HS, Lee DH. Change in Posterior Tibial Slope After Open-Wedge and Closed-Wedge High Tibial Osteotomy: A Meta-analysis. Am J Sports Med. 2016 Nov;44(11):3006-3013. doi: 10.1177/0363546515626172. Epub 2016 Feb 12. PMID 26872893
- [Background] Noyes FR, Goebel SX, West J. Opening wedge tibial osteotomy: the 3-triangle method to correct axial alignment and tibial slope. Am J Sports Med. 2005 Mar;33(3):378-87. doi: 10.1177/0363546504269034. PMID 15716253
- [Background] Song KY, Koh IJ, Kim MS, Choi NY, Jeong JH, In Y. Early experience of lateral hinge fracture during medial opening-wedge high tibial osteotomy: incidence and clinical outcomes. Arch Orthop Trauma Surg. 2020 Feb;140(2):161-169. doi: 10.1007/s00402-019-03237-0. Epub 2019 Jul 4. PMID 31273455
- [Background] Teng Y, Mizu-Uchi H, Xia Y, Akasaki Y, Akiyama T, Kawahara S, Nakashima Y. Axial But Not Sagittal Hinge Axis Affects Posterior Tibial Slope in Medial Open-Wedge High Tibial Osteotomy: A 3-Dimensional Surgical Simulation Study. Arthroscopy. 2021 Jul;37(7):2191-2201. doi: 10.1016/j.arthro.2021.01.063. Epub 2021 Feb 11. PMID 33581296
- [Background] Tischer T, Paul J, Pape D, Hirschmann MT, Imhoff AB, Hinterwimmer S, Feucht MJ. The Impact of Osseous Malalignment and Realignment Procedures in Knee Ligament Surgery: A Systematic Review of the Clinical Evidence. Orthop J Sports Med. 2017 Mar 27;5(3):2325967117697287. doi: 10.1177/2325967117697287. eCollection 2017 Mar. PMID 28451605
- [Background] Vadhera AS, Knapik DM, Gursoy S, Farivar D, Perry AK, Cole BJ, Chahla J. Current Concepts in Anterior Tibial Closing Wedge Osteotomies for Anterior Cruciate Ligament Deficient Knees. Curr Rev Musculoskelet Med. 2021 Dec;14(6):485-492. doi: 10.1007/s12178-021-09729-0. Epub 2021 Dec 15. PMID 34907514
- [Background] Won HH, Chang CB, Je MS, Chang MJ, Kim TK. Coronal limb alignment and indications for high tibial osteotomy in patients undergoing revision ACL reconstruction. Clin Orthop Relat Res. 2013 Nov;471(11):3504-11. doi: 10.1007/s11999-013-3185-2. Epub 2013 Jul 23. PMID 23877556
- [Background] Wu CC. Is clinical measurement of anatomic axis of the femur adequate? Acta Orthop. 2017 Aug;88(4):407-410. doi: 10.1080/17453674.2017.1304788. Epub 2017 Mar 23. PMID 28333575
- [Background] Yang JC, Chen CF, Luo CA, Chang MC, Lee OK, Huang Y, Lin SC. Clinical Experience Using a 3D-Printed Patient-Specific Instrument for Medial Opening Wedge High Tibial Osteotomy. Biomed Res Int. 2018 May 8;2018:9246529. doi: 10.1155/2018/9246529. eCollection 2018. PMID 29854810